CLINICAL TRIAL: NCT04388982
Title: Open-Label, Single-Center, Phase I/Ⅱ Clinical Trial to Evaluate the Safety and the Efficacy of Exosomes Derived From Allogenic Adipose Mesenchymal Stem Cells in Patients With Mild to Moderate Dementia Due to Alzheimer's Disease
Brief Title: the Safety and the Efficacy Evaluation of Allogenic Adipose MSC-Exos in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBMG-AD-01
Record Dates: First submitted 2020-04-28; First posted 2020-05-15 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSCs-Exos Dosage 1 (Experimental): MSCs-Exos. low-dose group
  Interventions: Biological: low dosage MSCs-Exos administrated for nasal drip
- MSCs-Exos Dosage 2 (Experimental): MSCs-Exos mid-dose group
  Interventions: Biological: mild dosage MSCs-Exos administrated for nasal drip
- MSCs-Exos Dosage 3 (Experimental): MSCs-Exos high-dose group
  Interventions: Biological: high dosage MSCs-Exos administrated for nasal drip

INTERVENTIONS:
Biological: low dosage MSCs-Exos administrated for nasal drip — Dosage：5μg MSCs-Exos,Total volume： 1ml Frequency：Twice a week Duration：12 weeks
  Arms: MSCs-Exos Dosage 1
Biological: mild dosage MSCs-Exos administrated for nasal drip — Dosage：10μg MSCs-Exos,Total volume： 1ml Frequency：Twice a week Duration：12 weeks
  Arms: MSCs-Exos Dosage 2
Biological: high dosage MSCs-Exos administrated for nasal drip — Dosage：20μg MSCs-Exos,Total volume： 1ml Frequency：Twice a week Duration：12 weeks
  Arms: MSCs-Exos Dosage 3

SUMMARY:
Evaluate the Safety and Efficacy of Exosomes Derived from Allogenic Adipose Mesenchymal Stem Cells（MSCs-Exos）in Subjects with Alzheimer's disease.

DETAILED DESCRIPTION:
To date, the main pathological characteristics of AD patients are the accumulation of β-amyloid (Aβ) into senile plaques, the abnormal aggregation of intracellular Tau protein to form neuron fiber tangles (NFT) and neuron death. There are still no effective treatments to prevent, halt, or reverse Alzheimer's disease.

Exosomes are naturally occurring nanosized vesicles and comprised of natural lipid bilayers with the abundance of adhesive proteins that readily interact with cellular membranes. These vesicles have a content that includes cytokines and growth factors, signaling lipids, mRNAs, and regulatory miRNAs. Exosomes are involved in cell-to-cell communication, cell signaling, and altering cell or tissue metabolism at short or long distances in the body, and can influence tissue responses to injury, infection, and disease.

The purpose of this single center, open label, phase I/Ⅱ clinical trial, therefore, is to explore the safety and efficacy of the exosomes derived from allogenic adipose mesenchymal stem cells (MSCs-Exos) in the treatment of mild to moderate dementia due to Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects themselves and their legal representatives (or their immediate family members) voluntarily received the treatment and signed the consent form before this study;
2. Age ≧ 50 years, males and females;
3. Subjects diagnosed with Patients with mild or moderate Alzheimer's disease, based on the NIA/AA(2011).
4. The Mini-Mental Status Examination (MMSE) score was 10-24 (inclusive);
5. Modified Hachinski Ischemic Scale (MHIS) score was ≦ 4;
6. Suspension of cognitive-enhancing drugs and marketed therapeutic drugs such as ginkgo, high-dose vitamin E, lecithin, estrogen, non-steroidal anti-inflammatory drugs (NSAIDs), Donepezil, Memantine, etc ;
7. Based on medical history, physical examination, vital signs, laboratory tests and 12-lead electrocardiogram (ECG) results, subjects are generally in good condition;
8. Subjects can walk independently or receive outpatient follow-up with assistive devices (wheelchairs, walkers or crutches), while the subject's vision and hearing (allowing glasses and / or hearing aids) do not affect the follow-up procedure;
9. The subject has an identified and reliable caregiver who must also meet the following conditions:

(1) In the hospital, caregiver can independently read and understand relevant research documents, and can do necessary communication with the investigator; (2) Caregiver can follow clinical research procedures and ensure that accurate information about the status of the subject can be provided during the study; (3) Caregiver live with the subject; or take care of the subject no less than 3 days a week and no less than 2 hours a day; 10. Female subjects with fertility (including women of childbearing age and women less than 1 year after menopause) were required to take effective contraception throughout the study. At the same time, urine pregnancy tests were negative during screening.

Exclusion Criteria:

1. The subjects with more serious allergic constitution;
2. Received allogeneic mesenchymal progenitor cell therapy or its derived exosomes;
3. Laboratory test (any item meets): neutrophil absolute number < 1.0 × 109 / L, platelet count < 100 × 109 / L, serum albumin < 30g / L, serum creatinine > upper limit of normal value range, total bilirubin, alanine aminotransferase, aspartate aminotransferase > upper limit of 2 times of normal value range;
4. The subject has serious and poorly controlled concomitant diseases, such as (but not limited to) cardiovascular, cerebrovascular, liver, kidney, lung, endocrine and other system diseases;
5. Severe Alzheimer's Disease;
6. Severe depression;
7. The subjects suffered from Parkinson's disease, multiple cerebral infarction, vascular dementia, Huntington's disease, hydrocephalus, progressive supranuclear paralysis, multiple sclerosis, epilepsy, mental retardation or major history of brain injury (with or without persistent neurological impairment) or known brain structural abnormalities;
8. The subject has an history malignant tumor；
9. The subject has severe generalized infectious diseases in the 3 months prior to this trial.;
10. The subject has contraindication of MRI, included but not only: the subject installed heart pacemaker, defibrillator, heart bracket, heart valve prosthesis, metal clip after aneurysm surgery, drug infusion device implanted in vivo, any electronic device implanted in the body (nerve stimulator, bone growth stimulator) endovascular coil, strainer, ECG monitor, metal suture, shrapnel or sand of body, plate fixation and steel nail after fracture surgery, artificial cochlea, middle ear shift plant, metallic intraocular foreign body etc; the subject is a claustrophobia, critical ill patient and so on.
11. The subject tests positive for: HIV, HBV, HCV and treponema pallidum;
12. The subject has history of alcoholism, drug abuse, or mental illness in the 10 years prior to this trial.
13. The subject has participated in any other clinical trial in the 6 months prior to this trial;
14. The female subjects are pregnant, lactating or pregnant in the past half a year;
15. The subject has any other unsuitable condition (such as factors reducing the follow-up compliance) to be determined by the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related abnormal laboratory values of Liver or kidney function | 12 weeks
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 weeks

SECONDARY OUTCOMES:
Cognitive function | baseline
  ADAS-cog (Alzheimer 's disease assessment scale-cognitive section) consists of 12 items. Maximum value is 70 and higher score means a worse congnitive condition.
Cognitive function | 12 weeks
  ADAS-cog (Alzheimer 's disease assessment scale-cognitive section) consists of 12 items. Maximum value is 70 and higher score means a worse congnitive condition.
Cognitive function | 24 weeks
  ADAS-cog (Alzheimer 's disease assessment scale-cognitive section) consists of 12 items. Maximum value is 70 and higher score means a worse congnitive condition.
Cognitive function | 36 weeks
  ADAS-cog (Alzheimer 's disease assessment scale-cognitive section) consists of 12 items. Maximum value is 70 and higher score means a worse congnitive condition.
Cognitive function | 48 weeks
  ADAS-cog (Alzheimer 's disease assessment scale-cognitive section) consists of 12 items. Maximum value is 70 and higher score means a worse congnitive condition.
Quality of life evaluation | baseline
  Scores of ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) range from 0 to 54 and higher score means a better life quality.
Quality of life evaluation | 12 weeks
  Scores of ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) range from 0 to 54 and higher score means a better life quality.
Quality of life evaluation | 24 weeks
  Scores of ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) range from 0 to 54 and higher score means a better life quality.
Quality of life evaluation | 36 weeks
  Scores of ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) range from 0 to 54 and higher score means a better life quality.
Quality of life evaluation | 48 weeks
  Scores of ADCS-ADL (Alzheimer's Disease Cooperative Study Activities of Daily Living) range from 0 to 54 and higher score means a better life quality.
MRI Neuroimaging | baseline
  Evaluation of MRI（Magnetic Resonance Imaging)
MRI Neuroimaging | 48 weeks
  Evaluation of MRI（Magnetic Resonance Imaging)
PET-CT Neuroimaging | baseline
  Evaluation of and PET-CT（Positron Emission Computed Tomography- Computed Tomography)
PET-CT Neuroimaging | 48 weeks
  Evaluation of and PET-CT（Positron Emission Computed Tomography- Computed Tomography)

OTHER OUTCOMES:
Changes of AD biomarkers | baseline and 48 weeks
  Changes of Aβ in serum and cerebrospinal fluid will be tested at baseline and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD,PhD, Principal Investigator — Ruijin Hospital; Xiaoling Gao, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Pala M, Yilmaz SG. Circular RNAs, miRNAs, and Exosomes: Their Roles and Importance in Amyloid-Beta and Tau Pathologies in Alzheimer's Disease. Neural Plast. 2025 Apr 8;2025:9581369. doi: 10.1155/np/9581369. eCollection 2025. PMID 40235521
- [Derived] Xie X, Song Q, Dai C, Cui S, Tang R, Li S, Chang J, Li P, Wang J, Li J, Gao C, Chen H, Chen S, Ren R, Gao X, Wang G. Clinical safety and efficacy of allogenic human adipose mesenchymal stromal cells-derived exosomes in patients with mild to moderate Alzheimer's disease: a phase I/II clinical trial. Gen Psychiatr. 2023 Oct 11;36(5):e101143. doi: 10.1136/gpsych-2023-101143. eCollection 2023. PMID 37859748